CLINICAL TRIAL: NCT03177356
Title: Immediate Implant Placement With Deproteinized Bovine Bone (Tutogen) Versus Placement of Platelet-rich Fibrin as a Space Filling Material in Mandibular Molars. Randomized Clinical Trial.
Brief Title: Implant Placement in Mandibular Molar Xenograft Versus PRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hussein El Garhy, DR., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cebc.cairouniversity
Record Dates: First submitted 2017-06-03; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Platelet rich fibrin,xenograft

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extraction,implant placement,PRF (Experimental): Extraction of Mandibular first molar and Implant placement followed by Placement of placement of Platelet rich fibrin as space filling material
  Interventions: Procedure: extraction,implant placement,PRF
- Exctraction,Implant placement,Bone graft (Active Comparator): Extraction of mandibular first molar followed by implant placement and xenogenic bone graft as space filling material
  Interventions: Procedure: Exctraction,Implant placement,Bone graft

INTERVENTIONS:
Procedure: extraction,implant placement,PRF — Surgical extraction of mandibular molar using periotome and forceps followed by implant placement in inter-septal bone. Then a blood sample is withdrawn from patient and placed in the centrifuge. Then Platelet-Rich fibrin is placed in the extraction socket as space filling material
  Arms: extraction,implant placement,PRF
Procedure: Exctraction,Implant placement,Bone graft — Surgical extraction of mandibular molar using extraction forceps and periotome followed by implant placement in interseptal bone. De-proteinized bovine bone graft material is placed as space filling material
  Arms: Exctraction,Implant placement,Bone graft

SUMMARY:
20 recruited patients indicated for immediate implant placement in mandibular molar patients are divided into 2 groups each group contain 15 patients, one group assigned for placement of bovine bone after molar extraction and immediate implant placement, while the other group we use Platelet-rich fibrin as space filling material.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-restorable mandibular molars
2. Both sexes

   -

   Exclusion Criteria:
   * • Heavy smokers more than 20 cigarettes per day.5

     * Patients with in sufficient interseptal bone height and width

       * Patients with systemic disease that may affect normal healing.
       * Patients with completely resorbed buccal cortical plate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 1 week post operative
  evaluation of postoperative complications regarding pain and oedema

SECONDARY OUTCOMES:
implant stability | will be measure intraopertively immediately after insertion of the implants and will be measure one more time 6 months after 1st operation at the time of exposure of implants
  measurement of implant stability using osstell device
amount of bone gained or lost around the implants | 6 months postoperative
  two cone beam computed tomography (CBCT) will be taken for the patient, one immediate postoperative and the other 6 months after the operation then the height of bone gained or lost around the implants will be assessed by superimposing the same section in the two CBCTS

IPD SHARING:
Plan to Share IPD: Undecided